CLINICAL TRIAL: NCT07069569
Title: A Randomized, Open-Label, Multicenter Phase II Study to Evaluate the Efficacy and Safety of AHB-137 Injection in Combination With Hepatitis B Vaccine or Pegylated Interferon α-2b (Peg-IFN) in Participants With HBeAg-Negative Chronic Hepatitis B (CHB) Treated With Nucleos(t)Ide Analogue (NAs)
Brief Title: A Multicenter Study of AHB-137 Injection Combined With Other Hepatitis B Drugs
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ausper Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB-10-8007
Record Dates: First submitted 2025-06-25; First posted 2025-07-16 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AHB-137 (16 weeks) and Peg-IFN (Experimental)
  Interventions: Drug: AHB-137; Drug: Peg-IFN
- AHB-137 (24 weeks) and Peg-IFN (Experimental)
  Interventions: Drug: AHB-137; Drug: Peg-IFN
- AHB-137 and Hepatitis B vaccine (Experimental)
  Interventions: Drug: AHB-137; Drug: Hepatitis B Vaccine
- AHB-137 (Experimental)
  Interventions: Drug: AHB-137

INTERVENTIONS:
Drug: AHB-137 — AHB-137 will be injected.
Drug: Peg-IFN — Peg-IFN will be administered .
  Arms: AHB-137 (16 weeks) and Peg-IFN; AHB-137 (24 weeks) and Peg-IFN
Drug: Hepatitis B Vaccine — Hepatitis B vaccine will be administered.
  Arms: AHB-137 and Hepatitis B vaccine

SUMMARY:
This is a randomized, open-label, multicenter phase II study to evaluate the efficacy and safety of AHB-137 injection in combination with other hepatitis B drugs in participants with HBeAg-negative CHB treated with NAs.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily participate in the study, and sign the Informed Consent Form (ICF) prior to screening, able to complete the study according to the protocol;
* Aged between 18 and 65 years at the time of signing the ICF;
* Body mass index (BMI) within the range of 18-30 kg/ m2;
* HBeAg negative at screening;
* HBsAg or HBV DNA positive for at least 6 months;
* Continue antiviral therapy with a single nucleoside (t) ide analogue for more than 6 months prior to screening;
* Alanine aminotransferase (ALT) ≤ 2 × upper limit of normal (ULN);
* Effective contraception as required.

Exclusion Criteria:

* Participants who are not eligible for treatment with Peg-IFN/recombinant hepatitis B vaccine;
* Clinically significant abnormalities other than a history of chronic HBV infection;
* Concomitant clinically significant other liver diseases;
* Any serious infection other than chronic hepatitis B infection requiring intravenous anti-infective therapy within 1 month prior to screening;
* HCV RNA positive, Human immunodeficiency virus (HIV) positive, syphilis positive;
* Significant liver fibrosis or cirrhosis at screening, or a liver stiffness value (LSM) > 9.0 kPa;
* Previous/current manifestations of hepatic decompensation;
* Diagnosis or suspicion of hepatocellular carcinoma, or alpha-fetoprotein concentration (AFP) ≥ 20 ng/mL at screening;
* Obviously abnormal laboratory test results;
* History of vasculitis or presence of signs, symptoms, or laboratory tests of underlying vasculitis, and previous/current other diseases that may be related to vasculitic conditions;
* QT interval corrected for heart rate (Fridericia method) abnormal;
* History of extrahepatic disease possibly related to HBV immune status;
* Participants with a history of malignancy within the past 5 years or who are being evaluated for a possible malignancy;
* Serious mental illness or history of serious mental illness prior to screening;
* Suspected history of allergy to any component of the study drug, or allergic constitution;
* Major trauma or major surgery within 3 months prior to screening, or planned surgery during the study;
* Those who are participating in another clinical trial, or have not undergone a protocol-specified washout period prior to this study;
* Current use or use of any immunosuppressive medication within 3 months prior to screening, with the exception of short courses (≤ 2 weeks) or use of topical/inhaled steroids;Those who have used immunomodulators and cytotoxic drugs within 6 months prior to the first dose;Or a history of vaccination within 6 months prior to screening or a live vaccination plan during the trial;
* Participants requiring regular long-term administration of anticoagulants or antiplatelet drugs;
* Thyroid dysfunction;
* Patients with uncontrolled epilepsy and other progressive neurological disorders;
* Received any antisense oligonucleotides (ASO) or small molecule interfering ribonucleic acid (siRNA) drug;
* Any other circumstance or condition that, in the opinion of the investigator, the participants are inappropriate for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with persistent HBsAg < limit of detection (LOD) and HBV DNA < lower limit of quantification (LLOQ) at the 24th week after all treatment for CHB was discontinued. | up to 72 weeks

SECONDARY OUTCOMES:
Proportion of participants with persistent HBsAg < LOD and HBV DNA < LLOQ . | Up to 72 weeks
Detection of the serum concentration of HBsAg, HBsAb, HBV DNA, HBV RNA, HBcrAg, HBeAb,and HBeAg. | Up to 72 weeks
Proportion of participants who met discontinuation criteria for NAs treatment at the end of the treatment period. | Up to 48 weeks
Relapse rate after discontinuation of NAs therapy. | Up to 72 weeks
Change from baseline in alanine aminotransferase (ALT) values and time to normalization of values. | Up to 72 weeks
Relapse time after discontinuation of NAs therapy. | Up to 72 weeks
Plasma concentrations of AHB-137. | Up to 48 weeks
Serum concentrations of Peg-IFN. | Up to 48 weeks.
Safety: Number and percentage of participants with detectable anti-drug antibodies (ADA). | Up to 72 weeks
Safety: Changes of the hepatitis B quality of life (HBQOL) instrument in participants compared with baseline. | Up to 72 weeks
  This scale has 31 items, including 7 dimensions: psychological status, expected anxiety, vitality, shame, infectivity, health vulnerability, and viral response. Each item is scored on a 5-point scale, with higher scores indicating a more severe impact of hepatitis B on quality of life.
Safety: Number of participants with treatment-emergent adverse events (TEAEs), serious adverse events (SAE) and clinically significant examination results. | Up to 72 weeks
  Examination including laboratory examination, electrocardiogram (ECG) examination.
Safety: Monitoring the score changes of Columbia Suicide Severity Scale (CSSRS) . | Up to 72 weeks.
  The CSSRS is a categorical, interviewer-rated instrument that screens for suicidal ideation (five items, 0-1 each) and suicidal behavior (six items, 0-1 each); the highest positive item defines the risk level rather than a total score. For ideation items 3-5 an additional 0-5 intensity rating can be recorded. Across all items the minimum value is 0 (absent) and the maximum is 1 (present); a score of 1 on any item indicates a worse outcome and triggers escalating clinical safeguards, with any behavior item being tantamount to a suicidal event.
Safety: Changes of the score of EuroQol Five-Dimension Five-Level Scale (EQ-5D-5L) in participants compared with baseline. | Up to 72 weeks
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Safety: Monitoring the score changes of Self-Rating Depression Scale (SDS). | Up to 72 weeks.
  The SDS is a 20-item, 4-point Likert self-report scale that yields a raw sum of 20-80 points, conventionally converted to a standard score of 25-100 by multiplying the raw total by 1.25. Higher standard scores denote worse outcomes: <50 normal, 50-59 mild, 60-69 moderate, and ≥70 severe depression, with ≥70 warranting specialist evaluation and suicide-risk assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jia, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No